CLINICAL TRIAL: NCT05474898
Title: Magnesium Sulphate Iontophoresis Versus High- Power Pain Threshold Ultrasound in Mechanical Neck Pain
Brief Title: IONTOPHORESIS Versus Ultrasound in Mechanical Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hend Hamdy, lecturer of pt for basic science department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: p.T.RCE/012/003552
Record Dates: First submitted 2022-07-23; First posted 2022-07-26 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Trigger Point Pain, Myofascial
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (A) (Experimental)
  Interventions: Other: Magnesium Sulphate Iontophoresis +conventional therapy; Other: conventional theapy
- Group (B) (Experimental)
  Interventions: Other: High- Power Pain Threshold Ultrasound +conventional therapy; Other: conventional theapy
- Group (c) (Other)
  Interventions: Other: conventional theapy

INTERVENTIONS:
Other: Magnesium Sulphate Iontophoresis +conventional therapy — will receive Mgso4 Iontophoresis in addition to conventional therapy twice a week/4 weeks
  Arms: Group (A)
Other: High- Power Pain Threshold Ultrasound +conventional therapy — will receive HPPT-US on the upper trapezius in addition to conventional therapy twice a week/4 weeks
  Arms: Group (B)
Other: conventional theapy — will receive postural correction exercise-stretching and strengthening twice a week/4weeks

SUMMARY:
to investigate the effects of Magnesium Sulphate Iontophoresis versus High Power Pain Threshold Ultrasound on pain, function and range of motion on active MTrPs found in the upper trapezius.

DETAILED DESCRIPTION:
Myofascial pain syndrome (MPS) is a musculoskeletal chronic pain disorder that affects the majority of pain population and characterized by the presence of trigger points. MPS is usually associated with tenderness, spasm, movement limitation and referred pain .

Myofascial trigger points (MTrPs) are hyperirritable taut fibers of skeletal muscle. The taut fibers within the muscle create palpable nodules that may cause local pain, and refer pain elsewhere with soft tissue examination .

ELIGIBILITY:
Inclusion Criteria:

* Subjects, with age ranged from 19-23 years (Forman et al, 2014) from both genders. The subjects had active MTrPs in the upper fibers of trapezius muscle.

Exclusion Criteria:

* • History of whiplash injury.

  * History of cervical spine surgery.
  * Cervical radiculopathy or myelopathy.
  * Having undergone physical therapy within the past three months before the study.
  * Non- rheumatologic diseases as multiple sclerosis, thyroid dysfunction and chronic infection.
  * Rheumatologic condition as poly-articular osteoarthritis, rheumatoid arthritis and advanced cervical spine degenerative diseases.

Ages: 19 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
pain intensity | up to four weeks
  The scale that will be used the VAS ;each subject will instructed to put point on line from no pain to tolerable pain

SECONDARY OUTCOMES:
Pain pressure threshold (PPT) | up to four weeks
  Pain pressure threshold (PPT) is used to measure deep muscular tissue sensitivity by Algometer.
neck disability | up to four weeks
  will be measured by Arabic neck disability index
range of motion | up to four weeks
  will be measured by myrin gravity reference goniometer

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ibrahim NA, Hamdy HA, Elbanna RHM, Mohamed DMA, Ali EA. Transdermal iontophoresis versus high power pain threshold ultrasound in Mechanical Neck Pain: a randomized controlled trial. J Orthop Surg Res. 2024 Oct 15;19(1):658. doi: 10.1186/s13018-024-05078-z. PMID 39407315